CLINICAL TRIAL: NCT03918018
Title: SpO2 and Pulse Rate Accuracy Comparison of BiOSENCY BORA Band to Arterial Blood CO-Oximetry and Reference ECG
Brief Title: BiOSENCY BORA Band SpO2 Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosency (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PR2018-312
Record Dates: First submitted 2019-04-04; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hypoxia
Keywords: Pulse oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: BORA Band SpO2 Validation Study — Qualified healthy volunteers will be enrolled into the study. Subjects will recline for the study. Reference sensor(s) will be placed on each subject to evaluate the SpO2 accuracy and performance. Shield material may be used between any adjacent finger sensors to prevent optical crosstalk.
  Simultaneous data collection will be set up for device under test and the control pulse oximeter. The data from the test device will be collected by the sponsor or trained Clinimark Study staff. Data will be collected for 1 second intervals data analysis. The SpO2 accuracy of the test devices will be evaluated over the oxygen saturation range between 70-100%.
  The investigational device will only be placed on the wrist. The control pulse oximeter may be alternated through fingers between subjects.

SUMMARY:
The purpose of this clinical study is to validate the SpO2 accuracy of the BiOSENCY BORA BAND™ wristband Pulse Oximeter during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. The end goal is to provide supporting documentation for the SpO2 accuracy validation of BORA BAND™ wristband Pulse Oximeter.

It is required that the Accuracy Root Mean Square (ARMS) performance of the BORA BAND™ wristband Pulse Oximeter will meet a specification of 3.5 or better in non-motion conditions for the range of 70 - 100% SpO2 thereby demonstrating an acceptable SpO2 accuracy performance specification.

DETAILED DESCRIPTION:
The SpO2 accuracy performance of BiOSENCY BORA BAND™ wristband Pulse Oximeter will be evaluated during non-motion conditions over the range of 70-100% SaO2 and compared to arterial blood samples assessed by CO-Oximetry. A minimum of 10 healthy adult male and female subjects, ranging in age and pigmentation from light to dark, will be enrolled in the study to meet the study design requirements defined by ISO 80601-2-61:2017 and by the FDA's Guidance for Pulse Oximeters (March 4, 2013). The subjects will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels. The investigational device will be placed on the wrist opposite for the test per the instructions for use. Simultaneous data collection will be set up for the system under test and control oximeter.

For the data analysis, the control oximeter will be used to assess the stability of each data point. Data that is found to be unstable will be removed prior to the comparative analysis. The CO-Oximeter data will be reviewed to make sure it does not contain any anomalous values such as elevated, low or inconsistent COHb, MetHb, or tHb data. Anomalous values will be removed from the analysis prior to pairing of the SpO2 and SaO2 data. The statistical analysis is performed on a minimum of 200 data points collected from at least 10 subjects for the range of 70% to 100% SaO2 with allowance of ± 3% of the target range. Functional SaO2 as measured by Reference CO-Oximetry will be used as the basis for comparison. The Accuracy Root Mean Square (ARMS) calculation is used to determine the SpO2 accuracy performance. Success will be achieved with an ARMS of 3.5 or better showing equivalence to the Gold Standard Reference CO-Oximetry providing documentation to support SpO2 accuracy claims for the investigational device.

The study population will include 10-15 healthy non-smoking (or has refrained from smoking for 2 days) competent adults, 18-50 years of age. The subject selection will be an equitable distribution of males and females of any race with varying skin tones including at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger. The subjects must understand the study and consent to participate by signing the Informed Consent Form. The subjects must be healthy showing no evidence of medical problems as indicated by satisfactorily completing the health assessment form.

ELIGIBILITY:
Inclusion Criteria:

* 10-15 Adults with a minimum of 3 males and a minimum of 3 females, with the balance made up of either
* Subject must have the ability to understand and provide written informed consent
* Subject is 18 to 50 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study
* Wrist size should be between 15-23 cm (5.9 - 9 inches)

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, wrist, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Female subjects that are actively trying to get pregnant or are pregnant (confirmed by positive urine pregnancy test unless the subject is known to be not of child-bearing potential).
* Smoker Subjects who have refrained will be screened for COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Subjects with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery with continued indications of health issues ,
  * emphysema, COPD, lung disease
* Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings (reviewed during health screen).
  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent symptomatic head injury (within the last 2 months)
  * cancer / chemotherapy
* Subjects with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Subjects with severe allergies to iodine (only applicable if iodine is used)
* Subjects with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio < 0.4)
* Unwillingness or inability to remove colored nail polish from test digits.
* Other known health condition, should be considered upon disclosure in health assessment form
* Wrist size should be between 15-23 cm (5.9 - 9 inches)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Accuracy of BORA Band SpO2 measurements versus arterial blood co-oximetry | 1 day
  Accuracy of the BORA Band SpO2 measurement as compared to reference co-oximetry performed on arterial blood samples.
  Results shall include
  * SpO2 Root mean square accuracy of BORA Band
  * SpO2 Bias of BORA Band
  * Bland-Altman plots with linear regression line and 95% upper and lower limits of agreement
Accuracy of BORA Band Pulse Rate measurements versus electrocardiogram readings | 1 day
  Accuracy of the BORA Band pulse rate measurement as compared to reference electrocardiogram readings.
  Results shall include
  * Pulse rate Root mean square accuracy of BORA Band
  * Pulse rate Bias of BORA Band

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark Desaturation Laboratory, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT03918018/Prot_SAP_000.pdf